CLINICAL TRIAL: NCT03482700
Title: The Impact of Specialist Led Integrated Care on Guideline Adherence and Outcomes in COPD
Brief Title: Impact of Specialist Led Integrated Care in COPD
Acronym: INTEGR-COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Heart of England NHS Trust (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017069RM
Record Dates: First submitted 2018-02-16; First posted 2018-03-29 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: COPD
Keywords: COPD; GP Surgeries
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: There are two groups: An intervention group and a control group. The intervention group will have their usual annual COPD review performed by a specialist respiratory doctor at baseline and 12 months. The patients will receive care using our local COPD guidance which has been accepted by all local commissioning groups and secondary care organisations. The control group will receive the usual standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): The intervention group will have their usual annual COPD review performed by a specialist respiratory doctor at baseline and 12 months. The patients will receive care using our local COPD guidance which has been accepted by all local commissioning groups and secondary care organisations.
  Interventions: Behavioral: Intervention Arm
- Control (Other): Usual standard of care
  Interventions: Behavioral: Control Arm

INTERVENTIONS:
Behavioral: Intervention Arm — The intervention group will have their usual annual COPD review performed by a specialist respiratory doctor at baseline and 12 months. The patients will receive care using our local COPD guidance which has been accepted by all local commissioning groups and secondary care organisations.
  Arms: Intervention
Behavioral: Control Arm — Usual standard of care
  Arms: Control

SUMMARY:
This study will look at the impact of care delivery by a specialist respiratory doctor compared to general practitioners for patients with COPD in East Birmingham. The primary outcome will be to compare the rates of provision of guideline-based care in intervention and control practices.

DETAILED DESCRIPTION:
This study will look at the impact of care delivery by a specialist respiratory doctor compared to general practitioners for patients with COPD in East Birmingham. It will be run from the Heart of England NHS Foundation Trust, which will provide the specialist input and oversight, and up to 40 practices across the Eastern Birmingham Health Organisation with approximately 2200 patients with COPD confirmed by their current medical practitioner. Each practice will be randomised to either the intervention or control group. The intervention group will have their usual annual COPD review performed by a specialist respiratory doctor at baseline and 12 months. The patients will receive care using our local COPD guidance which has been accepted by all local commissioning groups and secondary care organisations. Treatment will be at the discretion of the clinician and is not specified in the trial protocol. The investigators anticipate that the treatment recommendations in the intervention arm may include referral to pulmonary rehabilitation and reduction in the use of inhaled corticosteroids, which are prescribed at high rates in our locality. The control group will be seen by the usual staff at their practice. These patients will not be seen by the trial team and their data will be extracted remotely using electronic systems.

The primary outcome will be to compare the rates of provision of guideline-based care in intervention and control practices. Secondary outcomes will include: referral to secondary care, unscheduled healthcare consultations (ED attendance, hospital admissions), COPD exacerbations, healthcare costs, medications prescribed, biochemical markers of disease, radiological investigations, lung function tests measured when clinically indicated, and death within 12 month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Practices will be eligible for inclusion if they give consent to data collection and are part of the EBHO.
* Patients from the practices will be eligible if they are coded to have COPD within the GP record. In addition patients who are not coded to have COPD in the GP record, but who have a hospital admission with a primary diagnosis of COPD within the enrolment period for practices (first 3 months) will be eligible.

Exclusion Criteria:

• Patients will only be excluded if they are proven not to have COPD at specialist assessment, or during the follow up period, as determined by changes in medical coding within the GP record. If patients are assessed by the specialist and the diagnosis is not felt to be robust, enrolment will be suspended until this matter can be clarified by use of post bronchodilator spirometry and/or other required parts of their clinical care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2017-12-06 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Rates of provision of guideline-based care in intervention and control practices for patients. | 1 Year
  This will be done via the number of patients concordant with local guidelines (where care is defined by medication received and non-pharmacological interventions received, and they must receive smoking cessation, pulmonary rehabilitation, self-management plan and appropriate COPD medications in order to be guideline compliant)

SECONDARY OUTCOMES:
Referral Outcome | 1 Year
  Referral to secondary care
Unscheduled Outcome | 1 Year
  Unscheduled healthcare consultations (ED attendance, hospital admissions)
COPD Outcomes | 1 Year
  COPD exacerbations
Healthcare Outcomes | 1 Year
  mean cost per patient in £ of the total cost of hospital attendances, GP visits, medications and vaccines during the study period
Medications Outcomes | 1 Year
  medications prescribed
Biochemical markers of disease Outcomes | 1 Year
  FBC, U&E, LFT, CRP, AAT level/phenotype, and sputum culture results taken for patient
Radiological Outcomes | 1 Year
  number of CT scans or Chest X rays done
Lung Function Outcomes | 1 Year
  Lung function tests measured when clinically indicated, FEV1 (l) and FEV1 (% predicted), FEV1/FVC
Death Outcome | 1 Year
  Death within 12 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Alice Turner, MD, Principal Investigator — Heart of England NHS Foundation Trust
Locations (1):
- Dr. Sarah Pountain, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No IPD plan

REFERENCES:
- [Derived] Patel K, Smith DJ, Huntley CC, Channa SD, Pye A, Dickens AP, Gale N, Turner AM. Exploring the causes of COPD misdiagnosis in primary care: A mixed methods study. PLoS One. 2024 Mar 6;19(3):e0298432. doi: 10.1371/journal.pone.0298432. eCollection 2024. PMID 38446828
- [Derived] Patel K, Pye A, Edgar RG, Beadle H, Ellis PR, Sitch A, Dickens AP, Turner AM. Cluster randomised controlled trial of specialist-led integrated COPD care (INTEGR COPD). Thorax. 2024 Feb 15;79(3):209-218. doi: 10.1136/thorax-2023-220435. PMID 38286619